CLINICAL TRIAL: NCT05071430
Title: Safety and Efficacy of HB-1 for Panic Disorder: A Multicenter, Randomized, Double Blind, Placebo-Controlled Trial
Brief Title: Safety and Efficacy of HB-1 for Panic Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Honeybrains Biotech LLC (Industry)
Collaborators: Cognitive Research Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HB-001
Record Dates: First submitted 2021-09-13; First posted 2021-10-08 (Actual); Results first posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-02

CONDITIONS: Panic Disorder
Keywords: panic; mental illness
MeSH Terms: conditions — Panic Disorder; Mental Disorders | interventions — Bulk Drugs

STUDY DESIGN:
Intervention Model Description: A sample size of 80 patients is planned for the study to be randomized in a 1:1 ratio of active to control.
Who Masked: Participant, Care Provider, Investigator
Masking Description: An unblinded pharmacist will be utilized to assign bottles to each patient using an Interactive Voice Response System (IVRS) central randomization system. Study treatment or placebo will be dispensed to patients in blinded bottles.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active Treatment (HB-01) (Active Comparator): Approximately 40 patients will receive HB-01 active study drug.
  Interventions: Drug: HB-01
- Placebo Treatment (Placebo Comparator): Approximately 40 patients will receive a matched placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HB-01 — HB-1 will be supplied as a dual active pharmaceutical ingredient tablet.
  Other Names: Active Drug
  Arms: Active Treatment (HB-01)
Drug: Placebo — HB-1 matched placebo
  Arms: Placebo Treatment

SUMMARY:
The purpose of this study is to determine the safety and efficacy of potential new treatment called "HB-1" versus placebo in male and female adult patients aged 18 to 60 years, inclusive, with panic disorder.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, placebo-controlled trial. All patients with panic disorder, with or without specified co-morbidities, who meet all of the inclusion and none of the exclusion criteria will be eligible. Patients and researchers will be blinded to their treatment group.

The study will enroll approximately 80 adult patients who meet the diagnosis of panic disorder.

The patients will be treated for 12 weeks including a 1 week safety follow up visit following the last dose of study drug.

ELIGIBILITY:
* Inclusion Criteria

  1. Male or female aged 18 to 60 years old, inclusive, at the time of informed consent.
  2. Meets Diagnostic and Statistical Manual of Mental Disorders (DSM-5) Criteria for Panic Disorder.
  3. Documented moderate to severe levels of symptoms at baseline (Panic Disorder Severity Scale of 13 or above)
  4. Medically stable on current medication regimen for at least 3 months including PRN ('as needed') medications as determined by Investigator.
  5. Willing to remain on current doses of other psychiatric medications throughout the length of the trial (unless a dose reduction is warranted due to improvement in symptoms).
  6. Willing and able to safely stop any of the following medications prior to study trial: Inhibitors or inducers of CYP3A4 (erythromycin, ritonavir, telithromycin, rifampin), HMG-CoA (hydroxy methylglutaric acid coagulase) Reductase Inhibitors (Simvastatin, Lovastatin, Atorvastatin), Beta Blockers (Timolol eyedrops, Metoprolol), Neuromuscular Blocking Agents (curare-like and depolarizing), Antihypertensive Agents (Prazosin and vasodilators, angiotensin-converting enzyme inhibitors, diuretics, beta blockers), Inhalation Anesthetics, Disopyramide, Flecainide, Quinidine, Cimetidine, Lithium, Carbamazepine, Phenobarbital, Cyclosporine, Digitalis, Aliskiren, Ramipril and Ramiprilat, aspirin.
  7. Fluent in English.
  8. Willing to take HB-1 or placebo.
  9. Willing and able to provide informed consent indicating an understanding of the requirements of the study and a willingness to comply with scheduled visits and all study procedures.
  10. Female patients must be surgically sterile (or have a monogamous partner who is surgically sterile) or be least 2 years postmenopausal or commits to use 2 acceptable forms of birth control (defined as the use of an intrauterine device, a barrier method with spermicide, condoms, any form of hormonal contraceptives, or abstinence) for the duration of the study and for 4 months following the last dose of study treatment. Male patients must be sterile (biologically or surgically) or commit to the use of a reliable method of birth control (condoms with spermicide) for the duration of the study and for 4 months following the last dose of study treatment. Individuals who are involved exclusively in same-sex relationships are exempt from the birth control requirements but must agree to abide by the recommendations if they do engage in a heterosexual relationship.
  11. Female patients who are women of childbearing potential (WOCBP) must have a negative pregnancy test at Screening, within 7 days of dosing with study treatment.
* Exclusion Criteria:

  1. Severe uncontrolled cardiac disease within 6 months of Screening, including but not limited to uncontrolled hypertension, hypotension (defined as below 90/60); unstable angina; myocardial infarction (MI) or cerebrovascular accident (CVA).
  2. Any clinically significant electrocardiogram (ECG) abnormalities at screening.
  3. Inadequate hepatic function defined as total bilirubin >1.5 × the upper limit of normal (ULN) ranges of each institution, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) >3 × the ULN range of each institution.
  4. Inadequate renal function defined as serum creatinine >1.5 × the ULN range of each institution and/or estimated glomerular filtration rate (eGFR) <60.
  5. Any clinically significant abnormalities in clinical laboratory assessments as assessed by the Investigator.
  6. Any other systemic conditions or organ abnormalities that in the opinion of the Investigator may interfere with the conduct and/or interpretation of the current study.
  7. Unable to complete neuropsychological testing.
  8. Diagnosis of Bipolar I, Bipolar II disorder or Schizophrenia.
  9. History of suicidal behaviors including ideation.
  10. Current treatment with doses of benzodiazepines that are outside the FDA-approved prescriber's information.
  11. Already on treatment with either telmisartan or verapamil or both.
  12. Documented prior drug allergy to either telmisartan or verapamil.
  13. Documented contraindication to taking telmisartan or verapamil: (eg, Duchenne's muscular dystrophy, myasthenia gravis).
  14. Documented moderate to severe substance abuse within the last 6 months (recreational cannabis use is allowed).
  15. Pregnant or breastfeeding.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 86 (Actual)
Dates: Start 2022-02-03 (Actual); Primary Completion 2022-12-12 (Actual); Study Completion 2022-12-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Walling, Principal Investigator — Collaborative NeuroScience Research, Garden Grove, CA
Locations (10):
- United States (10):
  - Collaborative Neuroscience Research, Garden Grove, California
  - Lumos Psychiatric Services, San Jose, California
  - Institute of Living, Hartford, Connecticut
  - CNS Healthcare, Jacksonville, Florida
  - CNS Healthcare, Orlando, Florida
  - Uptown Research Institute, Chicago, Illinois
  - Hassman Research Institute, Berlin, New Jersey
  - SPRI Clinical Trials, Brooklyn, New York
  - Richmond Behavioral Associates, Staten Island, New York
  - CNS Healthcare, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Three participants withdrew prior to receiving study treatment changing 86 to 83 subjects treated.
Groups:
- Active Treatment (HB-01): 42 patients received HB-01 active study drug.
  HB-01: HB-1 will be supplied as a dual active pharmaceutical ingredient tablet.
- Placebo Treatment: 41 patients received matched placebo.
  Placebo: HB-1 matched placebo
Period: Overall Study
Arm/Group | Active Treatment (HB-01) | Placebo Treatment
Started | 42 | 41
Completed | 32 | 32
Not Completed | 10 | 9
Not completed — Adverse Event | 1 | 2
Not completed — Lost to Follow-up | 4 | 4
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Other | 1 | 1

BASELINE CHARACTERISTICS:
Population: Of the 135 subjects screened, 86 subjects were randomized to the study, 44 to the treated group and 42 to the placebo group. 83 subjects received at least one dose of study medication, 42 in the active treatment arm and 41 in the placebo arm. Three participants withdrew prior to receiving study treatment.
Groups:
- Active Treatment (HB-01): 44 patients received HB-01 active study drug.
  HB-01: HB-1 will be supplied as a dual active pharmaceutical ingredient tablet.
- Placebo Treatment: Approximately 42 patients received matched placebo.
  Placebo: HB-1 matched placebo
- Total: Total of all reporting groups
Arm/Group | Active Treatment (HB-01) | Placebo Treatment | Total
Number analyzed (Participants) | 42 | 41 | 83
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 42 | 41 | 83
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.4 (10.25) | 36.3 (13.54) | 37.3 (11.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 30 | 61
  Male | 11 | 11 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 12 | 9 | 21
  White | 26 | 25 | 51
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 42 | 41 | 83

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Treatment-Emergent Adverse Events
Description: Safety was evaluated through Adverse Event monitoring, review of clinically significant changes in routine laboratory tests, ECGs, and orthostatic vital signs. The safety results were presented as: number of subjects reporting an adverse event as percentage of study population that met the eligibility criteria.
Time Frame: Up to 12 weeks
Population: Safety Population - subjects who were randomized and received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Active Treatment (HB-01) | Placebo Treatment
Number analyzed (Participants) | 42 | 41
Participants | 23 | 15

2. Primary Outcome: Change in Panic Disorder Symptom Severity Scale (PDSS)
Description: Percentage of patients who achieved panic free status after 12 weeks"
Time Frame: Up to 12 weeks
Population: Panic Disorder Severity Scale Score (PDSS) Change from Baseline (ITT Population)
Measure: Count of Participants; unit: Participants
Groups:
- Placebo Treatment: 42 patients received matched placebo.
  Placebo: HB-1 matched placebo
Arm/Group | Active Treatment (HB-01) | Placebo Treatment
Number analyzed (Participants) | 44 | 42
Participants | 35 | 35

3. Primary Outcome: Change in Clinical Global Impression-Severity Scale (CGI-S)
Description: CGI-S is a 7 point scale where 1 indicates "normal, not at all ill" and 7 indicates "amongst the most extremely ill patients".
Time Frame: Up to 12 weeks
Population: 3 subjects withdrew before dosing: only 83 treated.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Treatment (HB-01) | Placebo Treatment
Number analyzed (Participants) | 42 | 41
score on a scale | 2.95 (1.053) | 3.33 (0,986)

4. Secondary Outcome: Number of Panic Attacks
Description: The proportion of all subjects achieving panic-free status at the end of the study.
Time Frame: Up to 12 weeks
Population: Panic Frequency in the Entire ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Active Treatment (HB-01) | Placebo Treatment
Number analyzed (Participants) | 42 | 42
Participants | 17 | 10

ADVERSE EVENTS:
Time Frame: Up to 12 weeks.
Groups:
- Placebo Treatment: 41 patients received a matched placebo.
  Placebo: HB-1 matched placebo
Arm/Group | Active Treatment (HB-01) | Placebo Treatment
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/41
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/41
Other Adverse Events (participants affected / at risk) | 23/42 | 15/41
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Active Treatment (HB-01) (N=42) | Placebo Treatment (N=41)
Headache (Nervous system disorders) | 0 | 3
dizziness (Nervous system disorders) | 2 | 0
lightheadedness (Nervous system disorders) | 1 | 1
migraine (Nervous system disorders) | 1 | 1
dizziness on standing (Nervous system disorders) | 1 | 0
Drowsiness (Nervous system disorders) | 1 | 0
menstrual migraine (Nervous system disorders) | 1 | 0
vestibular migraine (Nervous system disorders) | 1 | 0
covid-19 (Infections and infestations) | 3 | 2
common cold (Infections and infestations) | 1 | 0
gastroenteritis (Infections and infestations) | 1 | 0
sinus infection (Infections and infestations) | 1 | 0
skin infection (Infections and infestations) | 1 | 0
stomach virus (Infections and infestations) | 1 | 0
URTI (Infections and infestations) | 0 | 1
UTI (Infections and infestations) | 1 | 0
nausea (Gastrointestinal disorders) | 3 | 2
constipation (Gastrointestinal disorders) | 1 | 0
diarrhoea (Gastrointestinal disorders) | 1 | 0
food poisoning (Gastrointestinal disorders) | 0 | 1
tooth impacted (Gastrointestinal disorders) | 1 | 0
vomiting (Gastrointestinal disorders) | 0 | 1
insomnia (Psychiatric disorders) | 3 | 2
bipiolar disorder (Psychiatric disorders) | 0 | 1
nightmares (Psychiatric disorders) | 0 | 1
sleep disturbance (Psychiatric disorders) | 1 | 0
vivid dreams (Psychiatric disorders) | 1 | 0
orthostatic hypotension (Vascular disorders) | 4 | 4
fatigue (General disorders) | 3 | 0
flu-like symptoms (General disorders) | 1 | 0
increased creatinine clearance (Investigations) | 0 | 1
increased creatinine phosphokinase (Investigations) | 1 | 0
abnormal uterine bleeding (Reproductive system and breast disorders) | 0 | 1
uterine cramps (Reproductive system and breast disorders) | 0 | 1
seasonal allergy (Immune system disorders) | 1 | 0
back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
sensitive skin (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-12-02): https://cdn.clinicaltrials.gov/large-docs/30/NCT05071430/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-08): https://cdn.clinicaltrials.gov/large-docs/30/NCT05071430/SAP_001.pdf